CLINICAL TRIAL: NCT00595101
Title: A Phase 2, 28-Day Parallel-Group, Double-Masked, Dose Finding Study Comparing The Safety And Efficacy Of PF-03187207 To Latanoprost In Patients With Primary Open Angle Glaucoma Or Ocular Hypertension.
Brief Title: A Phase 2, Dose Finding Study of PF-03187207 in Patients With Primary Open Angle Glaucoma or Ocular Hypertension.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A9441003
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Results first posted 2020-08-27 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- PF-03187207 High Dose and Latanoprost Vehicle (Experimental): A single drop of each, once daily in study eye for 28 days
  Interventions: Drug: PF-03187207; Drug: Latanoprost Vehicle
- Latanoprost 0.005% and PF-03187207 Vehicle (Experimental): A single drop of each, once daily in study eye for 28 days
  Interventions: Drug: Latanoprost 0.005%; Drug: PF-03187207 Vehicle
- PF-03187207 Medium Dose and Latanoprost Vehicle (Experimental): A single drop of each, once daily in study eye for 28 days
  Interventions: Drug: PF-03187207; Drug: Latanoprost Vehicle
- PF-03187207 Low Dose and Latanoprost Vehicle (Experimental): A single drop of each, once daily in study eye for 28 days
  Interventions: Drug: PF-03187207; Drug: Latanoprost Vehicle

INTERVENTIONS:
Drug: PF-03187207
  Arms: PF-03187207 High Dose and Latanoprost Vehicle; PF-03187207 Low Dose and Latanoprost Vehicle; PF-03187207 Medium Dose and Latanoprost Vehicle
Drug: Latanoprost 0.005%
  Arms: Latanoprost 0.005% and PF-03187207 Vehicle
Drug: PF-03187207 Vehicle — One drop in study eye once daily for the first 28 days to all subjects, followed by 28 days in combination with PF-03187207.
  Arms: Latanoprost 0.005% and PF-03187207 Vehicle
Drug: Latanoprost Vehicle
  Arms: PF-03187207 High Dose and Latanoprost Vehicle; PF-03187207 Low Dose and Latanoprost Vehicle; PF-03187207 Medium Dose and Latanoprost Vehicle

SUMMARY:
To investigate dose response, safety and efficacy of PF-03187207 in patients with primary open-angle glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* Man or woman at least 20 years of age
* Diagnosis of primary open-angle glaucoma or ocular hypertension in one or both eyes.

Exclusion Criteria:

* Closed/barely open anterior chamber angle or a history of acute angle closure in either eye
* Contraindications to latanoprost and nitric oxide treatment
* Known latanoprost non-responders

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2007-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ken Harper, Study Director — Bausch & Lomb Incorporated
Locations (13):
- Japan (13):
  - Pfizer Investigational Site, Narashino, Chiba
  - Pfizer Investigational Site, Shimachi, Chiba
  - Pfizer Investigational Site, Kawasaki, Kanagawa
  - Pfizer Investigational Site, Kasukabe, Saitama
  - Pfizer Investigational Site, Fuji, Shizuoka
  - Pfizer Investigational Site, Mishima, Shizuoka
  - Pfizer Investigational Site, Susono, Shizuoka
  - Pfizer Investigational Site, Hachiōji, Tokyo
  - Pfizer Investigational Site, Hamura, Tokyo
  - Pfizer Investigational Site, Minato, Tokyo
  - Pfizer Investigational Site, Musashino, Tokyo
  - Pfizer Investigational Site, Setagaya City, Tokyo
  - Pfizer Investigational Site, Shizuoka

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-0318 0.006%: PF-0318 0.006% once daily in the evening
- PF-0318 0.024%: PF-0318 0.024% once daily in the evening
- PF-0318 0.04%: PF-0318 0.04% once daily in the evening
- 0.005% Latanoprost: 0.005% latanoprost once daily in the evening
Period: Overall Study
Arm/Group | PF-0318 0.006% | PF-0318 0.024% | PF-0318 0.04% | 0.005% Latanoprost
Started | 29 | 29 | 29 | 30
Completed | 29 | 28 | 29 | 30
Not Completed | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-0318 0.006% | PF-0318 0.024% | PF-0318 0.04% | 0.005% Latanoprost | Total
Number analyzed (Participants) | 29 | 29 | 29 | 30 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (12.2) | 60.9 (18.0) | 58.8 (15.1) | 60.0 (17.3) | 59.5 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 18 | 16 | 59
  Male | 16 | 17 | 11 | 14 | 58

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Mean Diurnal Intraocular Pressure (IOP) in the Study Eye on Day 28
Description: Intraocular pressure (IOP) was measured using a Goldmann applanation tonometer. Diurnal IOP, defined as the mean IOP over the day based on values obtained at 8 AM, 10 AM, 1 PM, and 4 PM, was calculated for each visit. Both eyes were tested, with the right eye preceding the left eye. The operator initially set the dial at 10 mmHg, then looked through the slit lamp and adjusted the dial to take the reading, and then recorded the results. The procedure was repeated on the same eye twice consecutively. If the measurements were within 2 mmHg or less of each other, the mean of the 2 readings was recorded as the IOP at that time point. If the 2 readings were more than 2 mmHg of each other, a third (consecutive) reading was taken and the median (middle) IOP was recorded as the IOP at that time point.
Time Frame: Baseline, 28 days
Population: The Per Protocol (PP) population consisted of all subjects in the intention to treat (ITT) population excluding those who made major protocol violations before completing the study. The PP population was considered as the primary analysis population of efficacy (primary and secondary endpoints) of the study.
Measure: Mean (Standard Deviation); unit: mmHg (milimeters of mercury)
Arm/Group | PF-0318 0.006% | PF-0318 0.024% | PF-0318 0.04% | 0.005% Latanoprost
Number analyzed (Participants) | 28 | 27 | 27 | 30
mmHg (milimeters of mercury) | -5.12 (2.55) | -5.94 (3.09) | -5.02 (2.03) | -5.25 (2.53)

2. Secondary Outcome: Change From Baseline in Mean Intraocular Pressure (IOP) at Specific Time Points on Day 14 and Day 28
Description: Intraocular pressure (IOP) was measured using a Goldmann applanation tonometer. Both eyes were tested, with the right eye preceding the left eye. The operator initially set the dial at 10 mmHg, then looked through the slit lamp and adjusted the dial to take the reading, and then recorded the results. The procedure was repeated on the same eye twice consecutively. If the measurements were within 2 mmHg or less of each other, the mean of the 2 readings was recorded as the IOP at that time point. If the 2 readings were more than 2 mmHg of each other, a third (consecutive) reading was taken and the median (middle) IOP was recorded as the IOP at that time point.
Time Frame: Baseline, Day 14, Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg (milimeters of mercury)
Arm/Group | PF-0318 0.006% | PF-0318 0.024% | PF-0318 0.04% | 0.005% Latanoprost
Number analyzed (Participants) | 28 | 27 | 27 | 30
mmHg (milimeters of mercury)
  Day 14, 9am | -5.20 (2.97) | -5.87 (3.21) | -4.35 (2.76) | -5.53 (2.53)
  Day 28, 9am | -5.63 (3.29) | -6.11 (3.82) | -5.19 (2.71) | -5.33 (2.66)
  Day 28, 11am | -5.61 (3.20) | -6.07 (3.31) | -5.46 (2.56) | -5.65 (2.80)
  Day 28, 2pm | -4.57 (2.77) | -5.28 (3.17) | -4.85 (2.11) | -5.27 (3.11)
  Day 28, 5pm | -4.68 (2.47) | -6.28 (3.56) | -4.57 (2.53) | -4.73 (2.93)

3. Secondary Outcome: Target IOP
Description: Percentage of participants with IOP of 18 mmHg or Lower, 16 mmHg or Lower, or 14 mmHg or Lower at Any Visit Through Day 28. Intraocular pressure (IOP) was measured using a Goldmann applanation tonometer. Both eyes were tested, with the right eye preceding the left eye. The operator initially set the dial at 10 mmHg, then looked through the slit lamp and adjusted the dial to take the reading, and then recorded the results. The procedure was repeated on the same eye twice consecutively. If the measurements were within 2 mmHg or less of each other, the mean of the 2 readings was recorded as the IOP at that time point. If the 2 readings were more than 2 mmHg of each other, a third (consecutive) reading was taken and the median (middle) IOP was recorded as the IOP at that time point.
Time Frame: Up to 28 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PF-0318 0.006% | PF-0318 0.024% | PF-0318 0.04% | 0.005% Latanoprost
Number analyzed (Participants) | 28 | 27 | 27 | 30
Participants
  18 mmHg or lower | 9 | 11 | 13 | 9
  16 mmHg or lower | 4 | 2 | 3 | 3
  14 mmHg or lower | 0 | 1 | 0 | 2

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | PF-0318 0.006% | PF-0318 0.024% | PF-0318 0.04% | 0.005% Latanoprost
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 2/29 | 3/29 | 5/29 | 2/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-0318 0.006% (N=29) | PF-0318 0.024% (N=29) | PF-0318 0.04% (N=29) | 0.005% Latanoprost (N=30)
Conjunctival hyperaemia (Eye disorders) | 0 | 3 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 1 | 2 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details